CLINICAL TRIAL: NCT00093847
Title: S-adenosyl Methionine (SAMe) Augmentation of Selective Serotonin Reuptake Inhibitors (SSRIs) for Treatment-Resistant Depression (TRD)
Brief Title: Optimizing the Effectiveness of Selective Serotonin Reuptake Inhibitors (SSRIs) in Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, George I. Papakostas, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23MH069629 (NIH); K23MH069629 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: Selective Serotonin Reuptake Inhibitors; S-adenosyl Methionine; SSRI; SAMe
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Oral SAMe Tosylate (Experimental): Participants receiving the oral SAMe tosylate
  Interventions: Drug: S-adenosyl methione (SAMe)
- 2 Oral Placebo Pill Twice Daily (Placebo Comparator): Participants receiving placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-adenosyl methione (SAMe) — Oral SAMe tosylate, up to 1600 mg per day for 6 weeks
  Other Names: Oral SAMe tosylate
  Arms: 1 Oral SAMe Tosylate
Drug: Placebo — Placebo to be taken daily for 6 weeks
  Other Names: Pill identical in appearance to drug but placebo
  Arms: 2 Oral Placebo Pill Twice Daily

SUMMARY:
This study will determine the effectiveness of adding S-adenosyl methionine to antidepressant drug treatment in reducing depressive symptoms in depressed people who have not responded to antidepressants alone.

DETAILED DESCRIPTION:
Some people with depression do not respond well to antidepressant treatment. S-adenosyl methionine (SAMe) is a naturally occurring compound that may have antidepressant effects. SAMe may also enhance the effectiveness of other antidepressants, such as selective serotonin reuptake inhibitors (SSRIs). This study will determine the effectiveness of oral SAMe in enhancing the effects of SSRIs in patients currently not responding to SSRI treatment.

This study will last 6 weeks. No follow-up visits will occur. Participants will be randomly assigned to add either oral SAMe or placebo to their existing SSRI regimen for 6 weeks. Depression scales and self-report questionnaires regarding depressive symptoms will be used to assess participants at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Major depressive disorder
* Use of an SSRI for at least 6 weeks prior to study entry with partial or no response

Exclusion Criteria:

* History of psychosis
* Allergy to SAMe
* Alcohol or drug abuse in the past 3 months prior to study entry

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2004-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George I. Papakostas, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Papakostas GI, Alpert JE, Fava M. S-adenosyl-methionine in depression: a comprehensive review of the literature. Curr Psychiatry Rep. 2003 Dec;5(6):460-6. doi: 10.1007/s11920-003-0085-2. PMID 14609501
- [Result] Papakostas GI, Mischoulon D, Shyu I, Alpert JE, Fava M. S-adenosyl methionine (SAMe) augmentation of serotonin reuptake inhibitors for antidepressant nonresponders with major depressive disorder: a double-blind, randomized clinical trial. Am J Psychiatry. 2010 Aug;167(8):942-8. doi: 10.1176/appi.ajp.2009.09081198. Epub 2010 Jul 1. PMID 20595412
- [Derived] Mischoulon D, Alpert JE, Arning E, Bottiglieri T, Fava M, Papakostas GI. Bioavailability of S-adenosyl methionine and impact on response in a randomized, double-blind, placebo-controlled trial in major depressive disorder. J Clin Psychiatry. 2012 Jun;73(6):843-8. doi: 10.4088/JCP.11m07139. Epub 2012 May 15. PMID 22687580
- [Derived] Dording CM, Mischoulon D, Shyu I, Alpert JE, Papakostas GI. SAMe and sexual functioning. Eur Psychiatry. 2012 Aug;27(6):451-4. doi: 10.1016/j.eurpsy.2011.01.003. Epub 2011 Mar 12. PMID 21398094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 outpatients with major depressive disorder who were partial- or non-responders to SSRI/SNRI therapy were enrolled in this trial conducted at Massachusetts General Hospital.
Pre-assignment Details: This was a randomzized (1:1) double-blind, placebo-controlled adjunct study of oral SAMe tosylate (target doses of 800mg PO BiD) to standard SSRI and SNRI antidepressants for patients with MDD.
Groups:
- Adjunct Oral SAMe Tosylate 800mg PO BiD: Participants receiving the oral SAMe tosylate
- Oral Adjunct Placebo: Participants receiving placebo
Period: Overall Study
Arm/Group | Adjunct Oral SAMe Tosylate 800mg PO BiD | Oral Adjunct Placebo
Started | 39 | 34
Completed | 31 | 24
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adjunct Oral SAMe Tosylate 800mg PO BiD | Oral Adjunct Placebo | Total
Number analyzed (Participants) | 39 | 34 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 6 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (14.1) | 48.5 (11.3) | 50.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 18 | 11 | 29
Region of Enrollment [Number; unit: participants]
  United States | 39 | 34 | 73

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Rating Scale Remission Rates
Description: The proportion of remitters for SAMe versus placebo was 46.1% versus 17.6%. Remission is defined as a final score of 7 or less on Hamilton Depression Rating Scale 17 item .
Time Frame: Measured at Week 6
Population: ITT LOCF
Measure: Number; unit: Percentage of Remitters HDRS17
Arm/Group | Adjunct Oral SAMe Tosylate 800mg PO BiD | Oral Adjunct Placebo
Number analyzed (Participants) | 39 | 34
Percentage of Remitters HDRS17 | 46.1 | 17.6

2. Secondary Outcome: HDRS17 Responders
Description: 35.8% versus 11.7%. Response is defined as a 50 percent or more score reduction on on Hamilton Depression Rating Scale 17 item .
Time Frame: Measured at Week 6
Population: ITT LOCF
Measure: Number; unit: Percentage of Responders HDRS17
Arm/Group | Adjunct Oral SAMe Tosylate 800mg PO BiD | Oral Adjunct Placebo
Number analyzed (Participants) | 39 | 34
Percentage of Responders HDRS17 | 35.8 | 11.7

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Adjunct Oral SAMe Tosylate 800mg PO BiD | Oral Adjunct Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/34
Other Adverse Events (participants affected / at risk) | 20/39 | 19/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adjunct Oral SAMe Tosylate 800mg PO BiD (N=39) | Oral Adjunct Placebo (N=34)
Diarrhea (Gastrointestinal disorders) | 7 (7) | 5 (5)
Upper gastrointestinal upset (Gastrointestinal disorders) | 14 (14) | 7 (7)
Insomnia (Nervous system disorders) | 4 (4) | 2 (2)
Somnolence and fatigue (Nervous system disorders) | 4 (4) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 2 (2)
Activation (Nervous system disorders) | 3 (3) | 4 (4)
Vivid dreams (Nervous system disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No